CLINICAL TRIAL: NCT05011084
Title: Randomized Control Trial of Combined Cryotherapy With Compression Versus Cryotherapy Alone After Orthopaedic Surgery
Brief Title: Combined Cryotherapy With Compression Versus Cryotherapy Alone After Orthopaedic Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ashley Bozzay, MD, Principal Investigator, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2020-0310
Record Dates: First submitted 2021-07-12; First posted 2021-08-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Cryotherapy Effect; Compression; Postoperative Pain Management
Keywords: Postoperative Pain Management; Opioid Epidemic; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Game Ready Cryotherapy with Compression Group (Experimental): Post-operative treatment will involve using a Game Ready ® unit
  Interventions: Device: Game Ready Cryotherapy with Compression Group
- Control Cryotherapy Group (Active Comparator): Post-operative treatment will involve using the standard of care cryotherapy (i.e., traditional ice packs without compression).
  Interventions: Other: Control Cryotherapy Group

INTERVENTIONS:
Device: Game Ready Cryotherapy with Compression Group — Instead of using the traditional ice-pack cryotherapy (without compression), patients randomized into this group will use the Game Ready device, which uses cryotherapy with compression, during their post-operative treatment care.
  Arms: Game Ready Cryotherapy with Compression Group
Other: Control Cryotherapy Group — Patients randomized to the control group will use the standard of care, which is using traditional cryotherapy (i.e., an ice pack without compression)
  Arms: Control Cryotherapy Group

SUMMARY:
Cryotherapy has been used to enhance recovery after orthopaedic surgery. Many devices are available but few can guarantee a temperature regulation during a prolonged time and therefore have been criticized. The arrival of new advanced cryotherapy devices made it possible to test the effect of prolonged cooling on rehabilitation after arthroscopic orthopaedic procedures.

DETAILED DESCRIPTION:
Opioids are most commonly administered for the treatment of pain and are among the most prescribed drugs in the United States (US). Between 2003 and 2011, opioid prescriptions increased from 149 million to 238 million [3,5,7,11]. In 2004, while constituting only 4.5% of the world's population, the US consumed 99% of the global supply of hydrocodone [3,11]. These trends resulted in the Centers for Disease Control and Prevention recognizing opioid abuse as an epidemic [2,11].

Pain management after orthopaedic arthroscopic procedures is mandatory regardless of the surgical technique. Cold therapy (cryotherapy) has been widely used for many years in the treatment of postoperative pain management in orthopaedic surgery and most studies have reported better pain scores and reduced drug consumptions [1,6,8]. Cryotherapy involves applying a cold device to the skin surrounding the injured soft tissues to reduce the intraarticular temperature. It reduces local blood flow by vasoconstriction, which in turn also reduces local inflammatory reaction, swelling, and heat experience. It also decreases the conduction of nerve signals potentially reducing pain transmission [14,15]. Several cryotherapy options are available: first generation cold therapy like crushed ice in a plastic bag, cold or gel packs; second-generation cold therapy with circulating ice water with or without compression; and third-generation advanced computer-assisted devices with continuous controlled cold therapy.

Cryotherapy is the standard of care in some countries and rarely is used in others [17]. Conflicting evidence regarding the value of this treatment from randomized trials may contribute to that practice disparity [16]. Raynor et al [8] showed that cryotherapy has a statistically significant benefit in postoperative pain control, while no improvement in postoperative range of motion or drainage was found. Cryotherapy with compression units are inexpensive, easy to use, have a high level of patient satisfaction, and are rarely associated with adverse events. Raynor et al [8] concluded cryotherapy may be justified in the postoperative management of knee surgery.

Postoperative cryotherapy with compression was proposed as a method of reducing pain and the inflammatory response in the early postoperative period after orthopaedic arthroscopic procedures. Previous study results are equivocal. Kraeutler et al [12] reported that there does not appear to be a significant benefit to use of cold compression over standard ice wraps in patients undergoing shoulder arthroscopy for rotator cuff repair or subacromial decompression. While Alfuth et al [13] concluded no recommendations can be made regarding the question whether cold compression therapy or cold therapy should be preferred immediately after arthroscopic surgery of the shoulder. Our goal is to analyze the analgesic efficacy of cryotherapy after shoulder, knee, and hip arthroscopic procedures using the Game Ready © which is a second generation cryotherapy with compression system. The investigators hypothesize this may decrease postoperative opioid usage as well as be more cost effective when compared to first generation cryotherapy (ice packs without compression) for medical healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Eligible for DEERS (Defense Enrollment Eligibility Reporting System - A system that enables uniformed service members & family members to receive health care through TRICARE)
* Fluent in speaking, reading, and understanding English
* Scheduled to receive one of the following procedures: Knee arthroscopy, Shoulder arthroscopy, or Hip arthroscopy

Exclusion Criteria:

* Unable to understand and/or provide written informed consent
* Presence of concurrent additional injuries (e.g., both a knee and hip injury). Participants can only have one injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Change in the Defense and Veterans Pain Rating Scale (DVPRS) before and after each cryotherapy session | Post-operative days 1-14
  Quick survey to assess pain level in the moment before and after each cryotherapy session.
  The DVPRS consists of a basic traffic-light color code. Green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10. The DVPRS also includes an additional visual tool: facial expressions that correspond with each number. The faces range from a full happy face representing a pain level of zero to a grimacing face representing a pain level of 10.
Defense and Veterans Pain Rating Scale (DVPRS) at wake up | Post-operative days 1-14
  Quick survey to assess pain level in the moment at the time of wake up.
  The DVPRS consists of a basic traffic-light color code. Green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10. The DVPRS also includes an additional visual tool: facial expressions that correspond with each number. The faces range from a full happy face representing a pain level of zero to a grimacing face representing a pain level of 10.
Defense and Veterans Pain Rating Scale (DVPRS) right before bed time | Post-operative days 1-14
  Quick survey to assess pain level in the moment at the time right before going to sleep.
  The DVPRS consists of a basic traffic-light color code. Green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10. The DVPRS also includes an additional visual tool: facial expressions that correspond with each number. The faces range from a full happy face representing a pain level of zero to a grimacing face representing a pain level of 10.
Cryotherapy Device Usage | Post-operative days 1-14
  Patients will maintain a Daily Therapy Log to document their usage of the assigned cryotherapy device.
Medication Consumption | Post-operative days 1-14
  Patients will maintain a daily Medication Log to record their consumption of pain medications.
Demographics Survey | Pre-operation (baseline)
  Prior to undergoing their arthroscopy, participants will complete a brief Demographics survey, which asks relevant medical and service history and demographic questions including: sex, race/ethnicity, year of birth, marital status, military affiliation, branch of service, military rank, occupational specialty, and employment status.
Change in the Single Assessment Numeric Evaluation (SANE) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  The SANE score is a validated patient reported outcome measure. It is a single question score that asks, "how would you rate your condition today as a percentage of normal (0% to 100% scale with 100% being normal)?" The SANE score is collected as standard of care.
Change in the Defense and Veterans Pain Rating Scale (DVPRS) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  The DVPRS consists of a basic traffic-light color code. Green represents mild pain with a scale ranging from 0-4; yellow represents moderate pain with a scale ranging from 5-6, and red represents severe pain with a scale ranging from 7-10. The DVPRS also includes an additional visual tool: facial expressions that correspond with each number. The faces range from a full happy face representing a pain level of zero to a grimacing face representing a pain level of 10.
  Four supplemental questions are included in the DVPRS to help identify how pain affects an individual's lifestyle. These questions also include a numerical scale that ranges from zero to 10 for each question. The four supplemental questions ask about pain pertaining to: daily activity during the past 24 hours, mood during the past 24 hours, sleep during the past 24 hours, stress during the past 24 hours
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  This patient reported outcome measures the outcome of patients with musculoskeletal disorders by assessing physical function through a grading scale of activities of daily living
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  This patient reported outcome measures the extent to which pain hinders an individual's engagement with physical, mental, cognitive, emotional, recreational, and social activities
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Depression (DEP) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  This patient reported outcome focuses on affective and cognitive manifestations of depression rather than somatic symptoms such as appetite, fatigue and sleep
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety (ANX) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  This patient reported outcome focuses on fear (e.g., worry, feelings of panic), anxious misery (e.g., dread), hyperarousal (e.g., tension, nervousness, restlessness), and somatic symptoms related to arousal (e.g., cardiovascular symptoms, dizziness)
Change in the Patient Reported Outcomes Measurement Information System (PROMIS) Sleep Interference (SI) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  This patient reported outcome measures self-reported alertness, sleepiness, tiredness, and functional impairments associated with sleep problems during waking hours within the past seven days
Change in the American Shoulder and Elbow Surgeons Standardized Shoulder Form (ASES) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is one pain scale worth 50 points and ten activities of daily living worth 50 points
Change in the International Knee Documentation Committee (IKDC) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee
Change in the Hip Disability and Osteoarthritis Outcome Score (HOOS) from before surgery to after surgery | Pre-operation (baseline) and then post-operation at 2 weeks, 6 weeks, 6 months, 12 months, and 24 months
  The hip disability and osteoarthritis outcome score (HOOS) is a questionnaire intended to be used to assess the patient's opinion about their hip and associated problems and to evaluate symptoms and functional limitations related to the hip during a therapeutic process

CONTACTS AND LOCATIONS:
Overall Officials: Ashley B Bozzay, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be shared with anyone. Only aggregate results will be shared publicly.

REFERENCES:
- [Background] Barber FA, McGuire DA, Click S. Continuous-flow cold therapy for outpatient anterior cruciate ligament reconstruction. Arthroscopy. 1998 Mar;14(2):130-5. doi: 10.1016/s0749-8063(98)70030-1. PMID 9531122
- [Background] Chakravarthy B, Shah S, Lotfipour S. Prescription drug monitoring programs and other interventions to combat prescription opioid abuse. West J Emerg Med. 2012 Nov;13(5):422-5. doi: 10.5811/westjem.2012.7.12936. PMID 23357954
- [Background] Kuehn BM. Opioid prescriptions soar: increase in legitimate use as well as abuse. JAMA. 2007 Jan 17;297(3):249-51. doi: 10.1001/jama.297.3.249. No abstract available. PMID 17227967
- [Background] Kumar K, Gulotta LV, Dines JS, Allen AA, Cheng J, Fields KG, YaDeau JT, Wu CL. Unused Opioid Pills After Outpatient Shoulder Surgeries Given Current Perioperative Prescribing Habits. Am J Sports Med. 2017 Mar;45(3):636-641. doi: 10.1177/0363546517693665. Epub 2017 Feb 9. PMID 28182507
- [Background] Manchikanti L, Helm S 2nd, Fellows B, Janata JW, Pampati V, Grider JS, Boswell MV. Opioid epidemic in the United States. Pain Physician. 2012 Jul;15(3 Suppl):ES9-38. PMID 22786464
- [Background] Morsi E. Continuous-flow cold therapy after total knee arthroplasty. J Arthroplasty. 2002 Sep;17(6):718-22. doi: 10.1054/arth.2002.33562. PMID 12216025
- [Background] Nelson AD, Camilleri M. Chronic opioid induced constipation in patients with nonmalignant pain: challenges and opportunities. Therap Adv Gastroenterol. 2015 Jul;8(4):206-20. doi: 10.1177/1756283X15578608. PMID 26136838
- [Background] Raynor MC, Pietrobon R, Guller U, Higgins LD. Cryotherapy after ACL reconstruction: a meta-analysis. J Knee Surg. 2005 Apr;18(2):123-9. doi: 10.1055/s-0030-1248169. PMID 15915833
- [Background] Schoenfeld AJ, Belmont PJ Jr, Blucher JA, Jiang W, Chaudhary MA, Koehlmoos T, Kang JD, Haider AH. Sustained Preoperative Opioid Use Is a Predictor of Continued Use Following Spine Surgery. J Bone Joint Surg Am. 2018 Jun 6;100(11):914-921. doi: 10.2106/JBJS.17.00862. PMID 29870441
- [Background] Scully RE, Schoenfeld AJ, Jiang W, Lipsitz S, Chaudhary MA, Learn PA, Koehlmoos T, Haider AH, Nguyen LL. Defining Optimal Length of Opioid Pain Medication Prescription After Common Surgical Procedures. JAMA Surg. 2018 Jan 1;153(1):37-43. doi: 10.1001/jamasurg.2017.3132. PMID 28973092
- [Background] Syed UAM, Aleem AW, Wowkanech C, Weekes D, Freedman M, Tjoumakaris F, Abboud JA, Austin LS. Neer Award 2018: the effect of preoperative education on opioid consumption in patients undergoing arthroscopic rotator cuff repair: a prospective, randomized clinical trial. J Shoulder Elbow Surg. 2018 Jun;27(6):962-967. doi: 10.1016/j.jse.2018.02.039. Epub 2018 Mar 26. PMID 29599038
- [Background] Kraeutler MJ, Reynolds KA, Long C, McCarty EC. Compressive cryotherapy versus ice-a prospective, randomized study on postoperative pain in patients undergoing arthroscopic rotator cuff repair or subacromial decompression. J Shoulder Elbow Surg. 2015 Jun;24(6):854-9. doi: 10.1016/j.jse.2015.02.004. Epub 2015 Mar 29. PMID 25825138
- [Background] Alfuth M, Strietzel M, Vogler T, Rosenbaum D, Liem D. Cold versus cold compression therapy after shoulder arthroscopy: a prospective randomized clinical trial. Knee Surg Sports Traumatol Arthrosc. 2016 Jul;24(7):2209-15. doi: 10.1007/s00167-015-3534-7. Epub 2015 Feb 13. PMID 25677503
- [Background] Algafly AA, George KP. The effect of cryotherapy on nerve conduction velocity, pain threshold and pain tolerance. Br J Sports Med. 2007 Jun;41(6):365-9; discussion 369. doi: 10.1136/bjsm.2006.031237. Epub 2007 Jan 15. PMID 17224445
- [Background] Kullenberg B, Ylipaa S, Soderlund K, Resch S. Postoperative cryotherapy after total knee arthroplasty: a prospective study of 86 patients. J Arthroplasty. 2006 Dec;21(8):1175-9. doi: 10.1016/j.arth.2006.02.159. PMID 17162178
- [Background] Adie S, Naylor JM, Harris IA. Cryotherapy after total knee arthroplasty a systematic review and meta-analysis of randomized controlled trials. J Arthroplasty. 2010 Aug;25(5):709-15. doi: 10.1016/j.arth.2009.07.010. Epub 2009 Sep 2. PMID 19729279
- [Background] Barry S, Wallace L, Lamb S. Cryotherapy after total knee replacement: a survey of current practice. Physiother Res Int. 2003;8(3):111-20. doi: 10.1002/pri.279. PMID 14533367

DOCUMENTS (1):
  • Informed Consent Form (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT05011084/ICF_001.pdf